CLINICAL TRIAL: NCT05425511
Title: WELL-being Improvement Following a SOphrology Intervention in Hospital Staff
Acronym: So-Well
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Clermont Auvergne (UCA) (Unknown); Centre National de la Recherche Scientifique, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AOI 2020 DUTHEIL; 2020-A03236-33 (Other: ANSM)
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2024-11

CONDITIONS: Stress Related Disorder; Sophrology; Neurolinguistic Programming
Keywords: stress; heart rate variability; well-being

STUDY DESIGN:
Intervention Model Description: We will recruit workers from hospitals who will be randomized in two groups:
  * the intervention group will have a longitudinal follow-up of seven months in total (a control period of 1 month, then 6 to 8 sophrology sessions during two months, then a 4-month follow-up)
  * the control group will have a differed intervention (longitudinal follow-up of seven months in total beginning by a control period without intervention of 3 months, then 6 to 8 sophrology sessions during two months, then a 2-month follow-up).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The intervention group will have a longitudinal follow-up of seven months in total (a control period of 1 month, then 6 to 8 sophrology sessions during two months, then a 4-month follow-up).
  Interventions: Behavioral: sophrology / neurolinguistic programming intervention
- control group (Active Comparator): The control group will have a differed intervention (longitudinal follow-up of seven months in total beginning by a control period without intervention of 3 months, then 6 to 8 sophrology sessions during two months, then a 2-month follow-up).
  Interventions: Behavioral: sophrology / neurolinguistic programming intervention

INTERVENTIONS:
Behavioral: sophrology / neurolinguistic programming intervention — 2 sessions will be offered per week at 2 different time and will last 1 hour. They can take place in a seated or standing position, without physical contact. The sessions will consist of breathing exercises, visualization, dynamic relaxation and concentration exercises. The program is standardized:
  1. Dialogue between the sophrologist and the participants. It is possible to specify the objective(s) of the session. The sophrologist can ask more specific questions to adapt the session.
  2. Presentation of the conduct of the session (possible variations) and instructions promoting autonomy
  3. Guided by the sophrologist, the goal is to help free yourself from tensions, to play down a situation that worries and finally to realize that we can deal with. Exercises are adapted to the difficulties encountered by the participants.
  4. Time for free expression after the practice to promote the integration of the technique while giving elements to the sophrologist to guide the future sessions.

SUMMARY:
Work stress and psychosocial risks are a major public health problem. Health-care workers (HCW) are particularly at risk. Moreover, non-HCW staff of hospitals can also be at risk, with working environment described as the main risk factor. The University Hospital (CHU) of Clermont-Ferrand is one of the 3 CHUs in France with more than 10% absenteeism, and the first CHU for duration of sick leave. The political orientations favor an approach to improve the quality of life at work.

Sophrology is a psychocorporal method used as a therapeutic technique or experienced as a philosophy of life. It is an exclusively verbal and non-tactile method. It combines a set of techniques that will act both on the body and on the mind through breathing exercises, muscle relaxation and mental imagery (or visualization). It allows to find a state of well-being and to activate all physical and psychological potential in order to acquire a better knowledge of oneself. NLP is a set of communication and self-transformation techniques that focuses on reactions rather than the origins of behaviors. NLP associated with sophrology proposes above all to mobilize the resources of the unconscious.

Neurolinguistic programming (NLP) strategies are effective in the improvement in mental (anxiety and depression), physical, and social health, both in the general population, in individuals with social/psychological problems or in patients, both in hospital settings or outside hospital. Similary, sophrology also demonstrated some benefits on symptoms of patients. However, these approaches have never been provided in the workplace for the benefits of workers at risk of stress-related disorders.

This protocol may permit improvements of stress-related outcomes. Putative short-term benefits: This protocol may incidentally detect cardiac disorders. Any abnormality discovered will not be covered by promotor's insurance (our exploratory study cannot lead to such event) and will be supported by health insurance.

In general, the investigators aim to demonstrate the effectiveness of a workplace sophrology / NLP intervention for HCW at risk of stress-related disorders. Stress and well-being will be the target of the intervention, and will be measured both in a subjective (questionnaire) and objective (biomarkers).

DETAILED DESCRIPTION:
Work stress and psychosocial risks are a major public health problem. Health-care workers (HCW) are particularly at risk. Moreover, non-HCW staff of hospitals can also be at risk, with working environment described as the main risk factor. The University Hospital (CHU) of Clermont-Ferrand is one of the 3 CHUs in France with more than 10% absenteeism, and the first CHU for duration of sick leave. The political orientations favor an approach to improve the quality of life at work.

Sophrology is a psychocorporal method used as a therapeutic technique or experienced as a philosophy of life. It is an exclusively verbal and non-tactile method. It combines a set of techniques that will act both on the body and on the mind through breathing exercises, muscle relaxation and mental imagery (or visualization). It allows to find a state of well-being and to activate all physical and psychological potential in order to acquire a better knowledge of oneself. NLP is a set of communication and self-transformation techniques that focuses on reactions rather than the origins of behaviors. NLP associated with sophrology proposes above all to mobilize the resources of the unconscious.

Neurolinguistic programming (NLP) strategies are effective in the improvement in mental (anxiety and depression), physical, and social health, both in the general population, in individuals with social/psychological problems or in patients, both in hospital settings or outside hospital. Similary, sophrology also demonstrated some benefits on symptoms of patients. However, these approaches have never been provided in the workplace for the benefits of workers at risk of stress-related disorders.

This project proposes to evaluate the effects of a NLP and sophrology intervention for HCW, at the workplace. The investigators aim to evaluate both subjective and objective measures of stress.

This protocol may permit improvements of stress-related outcomes. Putative short-term benefits: This protocol may incidentally detect cardiac disorders. Any abnormality discovered will not be covered by promotor's insurance (our exploratory study cannot lead to such event) and will be supported by health insurance.

In general, the investigators aim to demonstrate the effectiveness of a workplace sophrology / NLP intervention for HCW at risk of stress-related disorders. Stress and well-being will be the target of the intervention, and will be measured both in a subjective (questionnaire) and objective (biomarkers).

The main objective is to demonstrate an improved heart rate variability in the intervention group during the period between month 1 (M1) and M3 (sophrology sessions) of the intervention group in comparison with the same control period M1 to M3 of the "deferred intervention" group.

The secondary objectives are to study for the following comparisons ((i) within groups: comparisons between and M0 to M7 by randomization group and (ii) between groups: comparisons at M5 and then between M0 and M7):

* The effects of the intervention on mental, physical and social health.
* The long-term effects of the intervention.
* The relationships between the perception of work and mental, physical and social health.
* The factors of success of the intervention (personality and perception of work, attendance rate, quality of personal practice, etc.)
* The effects on other biomarkers of stress such as other measures of the activity of the autonomic nervous system, DHEAS, cortisol, etc.

The study will be proposed to workers of the University Hospital of Clermont-Ferrand (CHU)) using the mailing list of the staff. Volunteers will send an email with their contact to the address so-well@chu-clermontferrand.fr. A Clinical Research Assistant will contact them back and give them a first quick explanation of the study by phone, and will send them the information letter, so they can read it prior to the inclusion visit. Investigators will undergo the inclusion visits, either physically or by teleconsultation. Investigators will explain to each volunteer, in an exhaustive, clear and adapted manner, the research procedure, the potential benefit and the adverse effects taking into account their specificity (state of health, age, profession, habits and life projects, family environment, etc.) and will answer all questions. They can sign the consent form either during the consultation or later after a reflection period of 8 days. In this case or for teleconsultation, the two signed consent forms will be returned by post or internal mail to the investigator. The investigator will keep one form, and the second form with both signature (investigator and volunteer) will be given to the volunteer at the baseline measure. They will be informed of the possibility, once their consent has been given, to withdraw it at any time.

Statistical analysis will be performed using Stata software (v15, Stata-Corp, College Station, US). Categorical parameters will be described in terms of numbers and frequencies, whereas continuous variables will be expressed as mean and standard deviation or median and [inter-quartile range] according to statistical distribution. The normality will be studied using Shapiro-Wilk test. Graphic representations will be complete presentations of results.

Patients will be described and compared between groups at inclusion according to the following variables: compliance with eligibility criteria, epidemiological characteristics, clinical characteristics and characteristics of possible treatments. The baseline comparability of the two groups will be assessed on the main characteristics of the participants and potential factors associated with the primary outcome. A possible difference between the two groups on one of these characteristics will be determined according to clinical considerations and not solely statistical ones.

Intergroup comparisons will be systematically conducted (1) without adjustment and (2) by adjusting for factors whose distribution could be unbalanced between groups.

All statistical tests will be two-sided and p<0.05 will be considered significant. Most of analyses of the secondary evaluation criteria will be exploratory. As discussed by Feise, the adjustment of the type I error will not be systematically proposed, but case by case in view of clinical considerations and not only statistical.

This study aims to demonstrate an improved heart rate variability in the intervention group, in comparison with the control group. According to previous data, it seems reasonable to estimate that effect-size, for the primary analysis between M1 and M3, will be around 0.5 for HRV parameters (e.g. log(lf/hf), rmssd, sdnn, pnn50). To highlight such clinically relevant difference, 85 participants per randomized group will be needed for a two-sided type I error at 5%, a statistical power at 90%. Finally, it is proposed to include 100 patients per group to consider lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

* worker (HCW or NHCW) from a hospital,
* age between 18-65 years,
* with a stress greater than 50 on a visual analogue scale (VAS) of stress,
* person able to give an informed consent to participate in research and
* affiliated with a Social Security scheme

Exclusion Criteria:

* Psychiatric, cardiovascular (heart failure, arrhythmia, etc.), hepatic (liver failure, etc.), renal (kidney failure, etc.), or endocrinological diseases (diabetes, etc.) judged by the investigator to be incompatible with the study because they may interfere with the measurements
* Non-affiliated to a health insurance
* Protected persons (minors, pregnant women, breastfeeding women, guardianship, curatorship, deprived of freedoms, safeguard of justice)
* Refusal to participate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-03-08 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
heart rate variability (HRV) Description : Abrupt changes in HRV signals will be explored. Time Frame : During 34 hours in five different conditions | Once per session of sophrology (6 to 8 sessions) during the 2 months intervention
  HRV will be explored in time and frequency domains using Zephyr™ BioHarness™ BT.
heart rate variability (HRV) Description : Abrupt changes in HRV signals will be explored. Time Frame : During 34 hours in five different conditions | Once per month during 6 months
  HRV will be explored in time and frequency domains using Zephyr™ BioHarness™ BT.

SECONDARY OUTCOMES:
Skin conductance | Once per session of sophrology (6 to 8 sessions) during the 2 months intervention
  Measure using Wristband electrodes - Empatica E4
Skin conductance | Once per month during 6 months
  Measure using Wristband electrodes - Empatica E4
Demographics variables | Once at inclusion
  Measure of age, gender, qualification, personal status using a questionnaire
Clinical measurements (height) | Once at inclusion
  Measure of height using a questionnaire
Clinical measurements (weight) | Once at inclusion
  Measure of weight using a questionnaire
Psychology and quality of life (depression) | 5 times : Month 0, Month 1, Month 3, Month 5 and Month 7
  Measure of depression using HAD 7 items
Psychology and quality of life (anxiety) | 5 times : Month 0, Month 1, Month 3, Month 5 and Month 7
  Measure of anxiety using HAD 7 items
Psychology and quality of life (burn-out) | 5 times : Month 0, Month 1, Month 3, Month 5 and Month 7
  Measure of burn-out using Maslach Burn-Out Inventory
Psychology and quality of life (perception of work) | 5 times : Month 0, Month 1, Month 3, Month 5 and Month 7
  Measure of perception of work using Job Content Questionnaire of Karasek
Psychology and quality of life (alexithymia) | 5 times : Month 0, Month 1, Month 3, Month 5 and Month 7
  Measure of alexithymia using Toronto Alexithymia Scale (TAS-20)
Psychology and quality of life (VAS stress at home) | Once per week during the whole protocol (8 month)
  Measure of stress at home using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a worse outcome
Psychology and quality of life (VAS stress at work) | Once per week during the whole protocol (8 month)
  Measure of stress at work using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a worse outcome
Psychology and quality of life (VAS fatigue) | Once per week during the whole protocol (8 month)
  Measure of fatigue using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a worse outcome
Psychology and quality of life (VAS sleep quality) | Once per week during the whole protocol (8 month)
  Measure of sleep quality using visual analog scale of 100 mm ranging from 0 (Bad) ot 100 (Excellent). Higher scores mean a better outcome
Psychology and quality of life (VAS anxiety) | Once per week during the whole protocol (8 month)
  Measure of anxiety using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a worse outcome
Psychology and quality of life (VAS mood) | Once per week during the whole protocol (8 month)
  Measure of mood using visual analog scale of 100 mm ranging from 0 (Bad) ot 100 (Excellent). Higher scores mean a better outcome
Psychology and quality of life (VAS family support) | Once per week during the whole protocol (8 month)
  Measure of family support using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a better outcome
Psychology and quality of life (VAS hierarchy support) | Once per week during the whole protocol (8 month)
  Measure of hierarchy support using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a better outcome
Psychology and quality of life (VAS colleagues support) | Once per week during the whole protocol (8 month)
  Measure of colleagues support using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a better outcome
Psychology and quality of life (VAS burnout) | Once per week during the whole protocol (8 month)
  Measure of burnout using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a worse outcome
Psychology and quality of life (VAS job control) | Once per week during the whole protocol (8 month)
  Measure of job control using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a better outcome
Psychology and quality of life (VAS job demand) | Once per week during the whole protocol (8 month)
  Measure of job demand using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a worse outcome
Psychology and quality of life (VAS effort reward imbalance) | Once per week during the whole protocol (8 month)
  Measure of effort reward imbalance using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a better outcome
Lifestyle (coffee, tea and food intakes) | Once per week during the whole protocol (8 month)
  Measure of coffee, tea and food intakes using a questionnaire
Lifestyle (physical activity) | Once per session of sophrology (6 to 8 sessions) during the 2 months intervention
  Measure of physical activity using Recent Physical Activity Questionnaire (RAPQ)
Lifestyle (physical activity) | Once per month during 6 months
  Measure of physical activity using Recent Physical Activity Questionnaire (RAPQ)
Lifestyle (physical activity) | Once per week during the whole protocol (8 month)
  Measure of physical activity using questionnaire
Lifestyle (alcohol, tobacco, cannabis and medication) | Once per week during the whole protocol (8 month)
  Measure of consumption of alcohol, tobacco, cannabis and medication using questionnaire
Sophrology practice (number of sessions per week) | Once per week during the whole protocol (8 month)
  Measure of number of sessions per week using questionnaire
Stress before the last sophrology session | Once per session of sophrology (6 to 8 sessions) during the 2 months intervention
  Measure of stress before the last sophrology session using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a worse outcome
Stress after the last sophrology session | Once per session of sophrology (6 to 8 sessions) during the 2 months intervention
  Measure of stress after the last sophrology session using visual analog scale of 100 mm ranging from 0 (Minimum) ot 100 (Maximum). Higher scores mean a worse outcome
Allostatic load (cortisol) | Once per session of sophrology (6 to 8 sessions) during the 2 months intervention
  Measure of cortisol using saliva sampling (and deep-freezing)
Allostatic load (cortisol) | Once per month during 6 months
  Measure of cortisol using saliva sampling (and deep-freezing)
Allostatic load (DHEAS) | Once per session of sophrology (6 to 8 sessions) during the 2 months intervention
  Measure of DHEAS using saliva sampling (and deep-freezing)
Allostatic load (DHEAS) | Once per month during 6 months
  Measure of DHEAS using saliva sampling (and deep-freezing)
Allostatic load (leptin) | Once per session of sophrology (6 to 8 sessions) during the 2 months intervention
  Measure of leptin using saliva sampling (and deep-freezing)
Allostatic load (leptin) | Once per month during 6 months
  Measure of leptin using saliva sampling (and deep-freezing)
Allostatic load (ghrelin) | Once per session of sophrology (6 to 8 sessions) during the 2 months intervention
  Measure of ghrelin using saliva sampling (and deep-freezing)
Allostatic load (ghrelin) | Once per month during 6 months
  Measure of ghrelinusing saliva sampling (and deep-freezing)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Dutheil, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Dutheil F, Parreira LM, Pereira B, Baldet M, Marson F, Chabaud C, Blot M, Baker JS, Zak M, Vallet G, Magnon V, Clinchamps M, Altun S. SOphrology Intervention to Improve WELL-Being in Hospital Staff (SO-WELL): Protocol for a Randomized Controlled Trial Study. Int J Environ Res Public Health. 2023 Jan 9;20(2):1185. doi: 10.3390/ijerph20021185. PMID 36673939